## **Cover Page**

## Participation Consent Form

Study Title: Mirror Therapy and Treadmill Training for Patients with Chronic Stroke. A Pilot Randomised Controlled Trial

Document creation date: December 12th 2014

NCT number [not yet assigned].

Identifiers: [NCT ID not yet assigned]

## **Participation Consent Form**

## Mirror therapy and treadmill training for patients with chronic stroke: A pilot randomised controlled trial

- 1. I confirm that I have received a copy of the Information Sheet for the above study. I have read it and I understand it. I have received an explanation of the nature and purpose of the study and what my involvement will be.
- 2. I have had time to consider whether to take part in this study and I have had the opportunity to ask questions.
- 3. I understand that my participation is voluntary and that I can decide to opt out of the research at any time.
- 4. I understand that all information gathered about me during this study will be treated with full confidentiality.

| 5. I agree to take part i | n the above study. | |
|---------------------------|--------------------|---------------|
| Name of patient | <br>Date | <br>Signature |